CLINICAL TRIAL: NCT02085785
Title: Home-based Weight Loss Intervention for Individuals With Lower Extremity Amputation
Brief Title: Weight Loss Intervention for Individuals With Lower Extremity Amputation
Acronym: MOVE-LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F6982-Wa
Record Dates: First submitted 2014-01-17; First posted 2014-03-13 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Lower Extremity Amputation
Keywords: weight loss; exercise; home-based; lower extremity amputation; pilot study
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coached (Experimental): Participants randomized to the coached arm will receive the same educational and self-monitoring materials as the self-directed group. In addition, participants in the coached arm will receive 11 calls from a health coach and a single visit to their home by an exercise specialist.
  Interventions: Behavioral: Coached group
- Self-directed (Active Comparator): Participants randomized to the self-directed arm will receive the same educational and self-monitoring materials as the coached group, but no home visit and no coaching calls. They will be encouraged to make behavior changes on their own.
  Interventions: Behavioral: Self-directed control group
- Screened (Other): Individuals who were contacted to inform them about the study or who contacted study personnel to express an interest in participating. This group is presented in order to present statistics on feasibility regarding recruitment
  Interventions: Other: Screened only

INTERVENTIONS:
Behavioral: Coached group — Participants randomized to the coached arm will receive 1) education and self-monitoring materials [e.g., a booklet, calorie count book, pedometer, and scale (if they do not have one)], 2) a home visit by an exercise specialist, and 3) 11 telephone calls (over a 20-week period) by a health coach who will utilize motivational interviewing techniques to help the participant set eating and activity goals and trouble shoot problems when they occur
  Arms: Coached
Behavioral: Self-directed control group — Participants randomized to the self-directed control arm will receive the same educational and self-monitoring materials as the coached group [e.g., a booklet, calorie count book, pedometer, and scale (if they do not have one)], but no home visit and no coaching calls. They will be encouraged to make behavior changes on their own.
  Arms: Self-directed
Other: Screened only — Screened only - No intervention -- individuals who are contacted and/or screened for eligibility
  Arms: Screened

SUMMARY:
The purpose of this study is to pilot test a program to help overweight and obese individuals with a lower extremity amputation (LEA) lose weight and become more physically active. The investigators will randomize approximately 30 individuals to either a self-directed weight loss program (n=15) or a coached weight loss program (n=15). The primary purpose of this pilot study is to determine if a home-based weight loss/physical activity (PA) intervention is feasible in individuals with a LEA. MOVE-LEAP is a 20-week program that involves 11 phone calls from a health coach and a single home visit by a physical therapist.

This pilot study aims to:

1. test the feasibility of recruiting overweight/obese individuals with LEA into a randomized trial;
2. assess whether the intervention can be delivered with high fidelity, and
3. evaluate whether the intervention is acceptable to and safe as determined by participant feedback, participation and retention for outcome measures.

DETAILED DESCRIPTION:
Participants randomized to the intervention arm will receive (1) a home visit by an exercise specialist and (2) a 20-week telephone-delivered weight loss program, modeled on the VA's Telephone Lifestyle Coaching Program (MOVE!TLC). All participants (both the coached arm and self-directed arm) will be mailed a MOVE-LEAP packet [containing eating and physical activity logs, information on how to set weight loss goals, suggestions for physical activity/exercise, dietary guides, etc.), a MOVE-LEAP handout booklet, calories counting book, a pedometer, exercise digital versatile disc (DVD), and a flip-booklet with exercises ("Exercise Guide for Persons with Limb Loss"). A bathroom scale will be provided for participants who do not already own one.

Participants in the coached arm will receive a home visit by an exercise specialist. This visit will occur 1-3 weeks after randomization. The exercise specialist will assess the participant's capabilities and interest regarding physical activity as well as his/her home environment for physical activity. Since each participant may have different physical capabilities and limitations, the type and intensity of physical activity will be tailored to each participant's preferences and their home and neighborhood/community environment and resources. If the participant is interested in performing physical activity outside their home, study staff will provide them with information about community resources for physical activities.

Participants in the coached arm will receive 11 calls by a study health coach. During the phone calls (weekly initially and then every other week), the health coach will review progress and help the participant to set "SMART" goals (Specific, Measurable, Attainable, Relevant and Time-limited) and will use motivational interviewing techniques to help the participant achieve those goals. Motivational interviewing is a style of counseling meant to increase participant engagement through strategic use of open-ended questions, reflective listening and positive affirmations. The study staff will review the participant's progress on his or her goals and help him or her problem solve to resolve challenges and modify goals as needed. During each session, the coach will discuss an educational topic relating to weight loss. Written materials on each topic are included the booklet.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity amputation (including toes) for at least 1 year
* overweight or obese
* <60 minutes drive-time to VA Puget Sound Health Care System - Seattle campus, willing to be randomized
* provides written, informed consent
* able to perform some form of aerobic exercise (e.g., walking, bicycling, swimming)
* has telephone
* able to complete study assessments

Exclusion Criteria:

* Co-morbidities which may be contraindicated or indicate no potential benefit from weight loss or increasing physical activity
* unlikely to be able to adhere to study protocol and complete questionnaires and measurements reliably
* recent or current (last 6 months) participation in a weight loss program, including taking weight loss medications
* only uses motorized (non-manual) wheelchair

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson J. Littman, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Littman AJ, Haselkorn JK, Arterburn DE, Boyko EJ. Pilot randomized trial of a telephone-delivered physical activity and weight management intervention for individuals with lower extremity amputation. Disabil Health J. 2019 Jan;12(1):43-50. doi: 10.1016/j.dhjo.2018.08.002. Epub 2018 Aug 10. PMID 30115584

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 303 participants were contacted to recruit them into the study [VHA patient (n=237) and UWMC or Harborview patient (n=56)] and 10 individuals contacted study personnel expressing an interest in participating (n=313)
  15 participants were consented and enrolled, but 313 individuals will be assessed for the purpose of assessing feasibility
Groups:
- Self-directed: Participants randomized to the self-directed arm will receive the same educational and self-monitoring materials as the coached group, but no home visit and no coaching calls. They will be encouraged to make behavior changes on their own.
  Self-directed control group: Participants randomized to the self-directed arm will receive the same educational and self-monitoring materials as the coached group [e.g., a booklet, calorie count book, pedometer, and scale (if they do not have one)], but no home visit and no coaching calls. They will be encouraged to make behavior changes on their own.
Period: Overall Study
Arm/Group | Coached | Self-directed
Started | 7 | 8
Completed | 5 | 6
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Individuals who completed all baseline procedures including consent are included. Those who consented to participate but did not complete all baseline procedures are not included as baseline participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Coached | Self-directed | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.6) | 56.6 (10.7) | 56.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Individuals That Were Randomized of Those Contacted (Feasibility)
Description: Specific components include yield by method, recruitment rate, refusal rates and reasons
Time Frame: During recruitment (expected duration of 12-15 months)
Population: 313 individuals were assessed for this outcome measure. Note that the number analyzed are those that we contacted via a mailing or who contacted the study after seeing a study flyer.
Measure: Number; unit: participants
Groups:
- Overall Study Feasibility: Reporting of recruitment and eligibility for the targeted population
Arm/Group | Overall Study Feasibility
Number analyzed (Participants) | 313
participants | 15

2. Secondary Outcome: Feasibility - Retention
Description: Number of randomized individuals who complete baseline and study exit visit
Time Frame: Follow-up assessments (all participants) and during intervention (intervention group only) (weekly, for 20 weeks)
Measure: Number; unit: participants
Arm/Group | Coached | Self-directed
Number analyzed (Participants) | 7 | 8
participants | 5 | 6

3. Secondary Outcome: Acceptability
Description: Acceptability of intervention will be assessed via a brief satisfaction survey - % who would recommend the program to a friend
Time Frame: At follow-up assessment (20-weeks follow-up)
Population: Number who reported that they would recommend the program to a friend. Intervention assessment questionnaires were not linked to other study data, so we are unable to report study group information. The number analyzed are those who completed the 20-week follow-up measure.
Measure: Count of Participants; unit: Participants
Groups:
- Self-directed + Coached Combined: Intervention assessment questionnaires were not linked to other study data, so we are unable to report study group information
Arm/Group | Self-directed + Coached Combined
Number analyzed (Participants) | 9
Participants | 8

4. Secondary Outcome: Change in Weight
Description: Changes between baseline and 20-weeks later (end of intervention)
Time Frame: Baseline and follow-up assessment (20-weeks after randomization)
Population: Those who were not assessed at 20 weeks were assumed to have the same values as at baseline (last observation carried forward)
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Coached | Self-directed
Number analyzed (Participants) | 7 | 8
pounds | -7.3 [-16.0 to 1.5] | 1.3 [-2.8 to 5.3]

5. Secondary Outcome: Change in 6-minute Walk Distance
Description: Change in 6-minute walk distance (ft) from baseline to follow-up
Time Frame: Baseline and at follow-up assessment (20-weeks after randomization)
Population: Baseline carried forward if 20-week follow-up data not collected
Measure: Mean (95% Confidence Interval); unit: feet
Arm/Group | Coached | Self-directed
Number analyzed (Participants) | 7 | 8
feet | 185.4 [-31.9 to 402.8] | 43.2 [-69.1 to 155.4]

ADVERSE EVENTS:
Arm/Group | Coached | Self-directed
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes